CLINICAL TRIAL: NCT02372500
Title: Randomised Controlled Trial of Chewing Gum to Reduce Post Operative Ileus in Elective Colorectal Surgery
Brief Title: Trial of Chewing Gum to Reduce Post Operative Ileus in Elective Colorectal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Countess of Chester NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dale Vimalachandran, Consultant Colorectal Surgeon, Countess of Chester NHS Foundation Trust
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Surg050/14
Record Dates: First submitted 2015-02-09; First posted 2015-02-26 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Colorectal Cancer; Surgery
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chewing gum (Experimental): Patients will chew sugar free gum three times a day
  Interventions: Dietary Supplement: Chewing gum
- Control (No Intervention): Normal post operative care

INTERVENTIONS:
Dietary Supplement: Chewing gum — Sugar free chewing gum
  Arms: Chewing gum

SUMMARY:
It is unknown whether post operative chewing gum will reduce post operative ileus. This study is a randomised controlled trial that will determine whether chewing gum three times a day following surgery will reduce post operative ileus. Time to passage of flatus will be used to determine that incidence of ileus.

DETAILED DESCRIPTION:
Patients will be randomised to one of two arms, the experimental arm will be chewing gum and the control arm will be normal post operative care.

The primary endpoint is time to passage of flatus (defined as end of operation to first passage of flatus, in minutes).

The trial will be unblinded to patients and observers and has been powered to demonstrate a 15% reduction in passage to flatus (130 patients required)

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective colorectal surgery (open and laparoscopic), able to given informed consent

Exclusion Criteria:

* Emergency colorectal surgery, unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Bowel function (as assessed by questionnaire) | Minutes (end of surgery to first passage of flatus, measured up to 4 weeks)
  Time to passage of flatus

SECONDARY OUTCOMES:
Diet (as assessed by questionnaire) | Minutes (end of surgery to first solid food, assessed by patient questionnaire up to 4 weeks from randomisation)
  Time to tolerating full diet
Length of stay | Days (till successful discharge from secondary care to home or respite care measured up to first 31 days)
Post op nausea and vomiting score (as recorded by visual analogue scale) | Recorded daily for first 5 days
  Post op nausea and vomiting score (PONV)
Morbidity | Days (recorded up to 30 days and defined by Clavien-Dindo scale)
  Post operative morbidity

CONTACTS AND LOCATIONS:
Overall Officials: Dale Vimalachandran, MD FRCS, Study Director — Countess of Chester; Rachel Clifford, MRCS, Principal Investigator — Countess of Chester
Locations (1):
- Countess of Chester Hospital, Chester, Cheshire, United Kingdom